CLINICAL TRIAL: NCT05904379
Title: A Phase Ib/II Clinical Trial of AK112 and AK104 With or Without Chemotherapy in Advanced Non-small Cell Lung Cancer
Brief Title: AK112 and AK104 With or Without Chemotherapy in Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-208
Record Dates: First submitted 2023-05-17; First posted 2023-06-15 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Advanced Non-small-cell Lung Cancer
MeSH Terms: interventions — Carboplatin; Paclitaxel; Pemetrexed; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- AK112, AK104 dose 1 plus carboplatin and paclitaxel (Experimental)
  Interventions: Drug: AK112; Drug: AK104; Drug: Carboplatin; Drug: paclitaxel
- AK112, AK104 dose 1 plus carboplatin and pemetrexed (Experimental)
  Interventions: Drug: AK112; Drug: AK104; Drug: Carboplatin; Drug: pemetrexed
- AK112, AK104 dose 2 plus carboplatin and paclitaxel (Experimental)
  Interventions: Drug: AK112; Drug: AK104; Drug: Carboplatin; Drug: paclitaxel
- AK112, AK104 dose 2 plus carboplatin and pemetrexed (Experimental)
  Interventions: Drug: AK112; Drug: AK104; Drug: Carboplatin; Drug: pemetrexed
- AK112 plus AK104 (Experimental)
  Interventions: Drug: AK112; Drug: AK104
- AK112, AK104 plus docetaxel (Experimental)
  Interventions: Drug: AK112; Drug: AK104; Drug: Docetaxel
- docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: AK112 — Subjects receive AK112 intravenously.
  Arms: AK112 plus AK104; AK112, AK104 dose 1 plus carboplatin and paclitaxel; AK112, AK104 dose 1 plus carboplatin and pemetrexed; AK112, AK104 dose 2 plus carboplatin and paclitaxel; AK112, AK104 dose 2 plus carboplatin and pemetrexed; AK112, AK104 plus docetaxel
Drug: AK104 — Subjects receive AK104 intravenously.
  Arms: AK112 plus AK104; AK112, AK104 dose 1 plus carboplatin and paclitaxel; AK112, AK104 dose 1 plus carboplatin and pemetrexed; AK112, AK104 dose 2 plus carboplatin and paclitaxel; AK112, AK104 dose 2 plus carboplatin and pemetrexed; AK112, AK104 plus docetaxel
Drug: Carboplatin — Subjects receive carboplatin intravenously.
  Arms: AK112, AK104 dose 1 plus carboplatin and paclitaxel; AK112, AK104 dose 1 plus carboplatin and pemetrexed; AK112, AK104 dose 2 plus carboplatin and paclitaxel; AK112, AK104 dose 2 plus carboplatin and pemetrexed
Drug: paclitaxel — Subjects receive paclitaxel intravenously.
  Arms: AK112, AK104 dose 1 plus carboplatin and paclitaxel; AK112, AK104 dose 2 plus carboplatin and paclitaxel
Drug: pemetrexed — Subjects receive pemetrexed intravenously.
  Arms: AK112, AK104 dose 1 plus carboplatin and pemetrexed; AK112, AK104 dose 2 plus carboplatin and pemetrexed
Drug: Docetaxel — Subjects receive docetaxel intravenously.
  Arms: AK112, AK104 plus docetaxel; docetaxel

SUMMARY:
This trial is a Phase Ib/II study. All patients are stage IIIB/C (unsuitable for radical therapy) or IV non-small cell lung cancer(NSCLC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the safety and efficacy of AK112 and AK104 with or without chemotherapy in subjects with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of NSCLC.
* Has Stage IIIB/C or IV NSCLC (American Joint Committee on Cancer [AJCC 8th]).
* 18-75 years old (at the time consent is obtained).
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue.
* Has a life expectancy of at least 3 months.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as determined by the site study team.
* Has no EGFR-sensitive mutations or ALK gene translocations.
* Has adequate organ function.
* Has recovered from the effects of any prior radiotherapy or surgery.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Has any histologically small cell carcinoma component.
* Is currently participating in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment.
* Has undergone major surgery within 30 days of Study Day 1.
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has an active infection requiring systemic therapy.
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has a history of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to day 1 of study treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety reflected by AE | Up to 2 approximately years
  Safety will be reflected by AE, which is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
ORR per RECIST v1.1 | Up to 2 approximately years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.

SECONDARY OUTCOMES:
OS | Up to 2 approximately years
  Overall Survival (OS) is defined as the time from the start of treatment with AK112 until death due to any cause.
DoR per RECIST v1.1 | Up to 2 approximately years
  Duration of response (DoR) assessed according to RECIST v1.1.
DCR per RECIST v1.1 | Up to 2 approximately years
  Disease control rate (DCR) assessed according to RECIST v1.1.
TTR per RECIST v1.1 | Up to 2 approximately years
  Time to response (TTR) is defined as the time to response base on RECIST v1.1.
PFS per RECIST v1.1 | Up to 2 approximately years
  Progression-free survival (PFS) is defined as the time from the date of Initial administration till the first documentation of disease progression assessed by the investigator or death due to any cause (whichever occurs first).
AK112 serum concentration | Up to 2 approximately years
  The serum concentration of AK112 of individual subjects at different time points.
AK104 serum concentration | Up to 2 approximately years
  The serum concentration of AK104 of individual subjects at different time points.
ADA | Up to 2 approximately years
  Number of subjects with detectable anti-drug antibodies (ADA).
PD-L1 expression | Up to 2 approximately years
  The correlationship between PD-L1 expression and efficacy.
ctDNA | Up to 2 approximately years
  The correlationship between ctDNA detection and efficacy.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Shanghai Pulmonary Hospital, Shanghai